CLINICAL TRIAL: NCT01539018
Title: A Phase II Trial of Sorafenib Plus Tegafur-uracil (UFT) vs. Sorafenib as First Line Systemic Treatment for Patients With Advanced Stage HCC, Unresectable & Not Eligible for Local Ablation &/or TACE
Brief Title: Sorafenib Plus Tegafur-uracil (UFT) Versus Sorafenib as First Line Systemic Treatment for Patients With Advanced Stage HCC, Unresectable & Not Eligible for Local Ablation and/or TACE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After interim results data showed no evidence of a difference between both groups
Sponsor: Egyptian Society of Liver Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESLC1 (SADAT study)
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Sorafenib; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib alone. (Active Comparator): Sorafenib 400 mg p.o. twice daily until progression or intolerable toxicity alone.
  Interventions: Drug: Sorafenib
- sorafenib plus tegafur-uracil (Experimental): Sorafenib 400 mg p.o. twice daily continuously and UFT 125mg/m2 PO BID For 4 weeks and to be repeated on day 36 till progression or intolerance
  Interventions: Drug: sorafenib plus tegafur-uracil

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400 mg p.o. twice daily until progression or intolerable toxicity alone.
  Other Names: nexavar alone
  Arms: Sorafenib alone.
Drug: sorafenib plus tegafur-uracil — Sorafenib 400 mg p.o. twice daily until progression or intolerable toxicity and TEGAFUR-URACIL 125mg/m2 PO BID For 4 weeks and to be repeated on day 36 till progression or intolerance
  Other Names: nexavar plus UFT
  Arms: sorafenib plus tegafur-uracil

SUMMARY:
* Unlike the Asian and western regions, The vast majority of the Egyptian/Arabic Hepatocellular Carcinoma (HCC) patients are hepatitis C virus (HCV) associated.
* According to the SHARP study subgroup analysis, it seems that HCV associated HCC patients derive the max benefit of Sorafenib, the absolute gain between the Sorafenib arm & the placebo in m OS = 7 months, HR=0.58 (95% CI: 0.37-0.91).
* In spite of improvement in terms of overall survival (OS) and time to progression (TTP), in all studies where Sorafenib was compared to placebo, the Sorafenib arm was not accompanied by a significant volumetric reduction, and this may explains the lack of any symptomatic improvement (time to symptomatic progression (TTSP) almost identical)
* Reviewing the chemotherapy outcome, although there is no convincing evidence in survival benefit to patients with advanced HCC, however true shrinkage (reduction in tumor size), has been consistently reported although the magnitude of response is lacking consistency.

This indicates the need for coupling Sorafenib to a chemotherapeutic agent but:

* For patients with Hepatocellular Carcinoma, the toxicity profile of any chemotherapeutic agent of choice to be added to Sorafenib should be take in consideration
* The agent to be added to Sorafenib should be effective in terms of Tumor Shrinkage & with minimal toxicity regarding:
* Cardio-toxicity
* HFSR
* Diarrhea
* Hepato-toxicity
* Bone marrow suppression (although not relevant to the toxicity profile of Sorafenib, yet the HCC patients may have HCV related thrombocytopenia and variable degree of hypersplenism related pancytopenia)

Circulatory Overload (Hypertension) Why Tegafur-uracil (UFT)?

* Efficacy: For UFT, although the efficacy data in HCC are not as extensive as Doxorubicin, however in one phase II study UFT could improve survival when compared with conservative management.
* UFT Toxicity Profile:

In a phase III trial to asses the compare Efficacy & Safety of UFT with that of 5 FU in treatment of m CRC, Hematological toxicities were minimal (0% Grade ¾ leukopenia, neutropenia, febrile neutropenia, thrombocytopenia & was 3% for anemia), while the most commonly seen SE was grade I & II Diarrhea

•Accordingly UFT may be considered as a potential partner to Sorafenib in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* 1-The patient must provide written informed consent prior to enrollment into the study.

  2-The patient must be at least 18 years of age. 3-Patients must have histologically or cytologically confirmed or radiologically confirmed (according to AASLD criteria) advanced (unresectable, and/or metastatic) HCC not eligible for local ablation or TACE.

  4-Patients must have measurable disease according to RECIST criteria (at least one uni-dimensional lesion measurable by CT-scan or MRI) 5-Patients must have a life expectancy of at least 12 weeks 6-Patients must have an Eastern Co-operative Oncology Group (ECOG) performance status of 0 -2, Child-Pugh class A and only B7 7-Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/μl
  * Total bilirubin ≤ 1.5 times the upper limit of normal
  * ALT and AST < 5 x upper limit of normal
  * Alkaline phosphatase ≤ 5 x upper limit of normal
  * PT-INR/PTT < 1.5 x upper limit of normal
  * Serum creatinine < 1.5 x upper limit
  * Amylase and lipase < 1.5 X the upper limit of normal 8-For patients, who have had major surgery or injury, the wound must be completely healed prior to receiving sorafenib treatment (4 weeks).

    9-Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Men use adequate birth control for at least 3 months after the last administration of sorafenib

Exclusion Criteria:

Excluded medical conditions:

* History of cardiac disease: congestive heart failure > NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
* History of HIV infection
* Patients with Child-Pugh class C hepatic impairment
* Patients with Child-Pugh class B (except 7 ) hepatic impairment
* Active clinically serious infections (grade 2 NCI-CTC version 3.0)
* Symptomatic metastatic brain or meningeal tumors
* Patients with seizure disorder requiring medication (such as steroids or antiepileptics)
* History of organ allograft
* Patients with evidence or history of bleeding due to OV
* Patients undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma

Patients not fulfilling inclusion criteria.

Excluded therapies and medications, previous and concomitant:

* Prior systemic anticancer chemotherapy or immunotherapy or targeted therapy is not allowed before study entry.
* Hormonal therapy shouldn't be given within 2 weeks before study entry and is not allowed during the study.
* Patients who failed previous transcatheter arterial chemoembolism must have at least 4 weeks treatment free interval before entering the study
* Radiotherapy during study or within 3 weeks of start of study drug.
* Major surgery within 4 weeks of start of study
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
time to progression (TTP):recist criteria | one year

SECONDARY OUTCOMES:
progression free survival (PFS):recist criteria | one year
Time to symptomatic improvement:FHSI-8 questionnaire | one year
Quality of Life Using EQ-5D questionnaire. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abdelazim, MD/PhD, Study Chair — Cairo University; Hesham Atef, MD/PhD, Principal Investigator — Cairo University; Ashraf Abdelaziz, MD/PhD, Principal Investigator — Cairo University; Mohammed Shaker, MD/PhD, Principal Investigator — Ain Shams University; Imam Waked, MD/PhD, Principal Investigator — Monofeiya university; Heba Elzawahry, MD/PhD, Principal Investigator — Cairo university, national cancer institute; Mohammed Ezz alarab, MD/PhD, Principal Investigator — NTMRI; Omar Abdel-Rahman, M.D./M.Sc., Study Director — Ain Shams University
Locations (5):
- Egypt (5):
  - Ain shams university, Cairo
  - Cairo University Hospitals, Cairo
  - National cancer institute, Cairo
  - NHTMRI, Cairo
  - National Liver Institute, Monofeiya